CLINICAL TRIAL: NCT00203580
Title: A Randomized Trial of the Effect of Low-Molecular-Weight Heparin Versus Warfarin Sodium on the Mortality in the Long-Term Treatment of Proximal Deep Vein Thrombosis (Main LITE Study)
Brief Title: Trial of the Effect of Low-Molecular-Weight Heparin (LMWH) Versus Warfarin on Mortality in the Long-Term Treatment of Proximal Deep Vein Thrombosis (DVT) (Main LITE Study)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Calgary (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); LEO Pharma (Industry); Dupont Applied Biosciences (Industry)
Allocation: Randomized | Masking: None | Purpose: Treatment
Other Study IDs: 2736-1
Record Dates: First submitted 2005-09-12; First posted 2005-09-20 (Estimated); Last update posted 2007-02-09 (Estimated); Status verified 2005-09

CONDITIONS: Thrombosis; Thromboembolism; Venous Thrombosis
Keywords: venous thromboembolism; low-molecular-weight heparin
MeSH Terms: conditions — Thrombosis; Thromboembolism; Venous Thrombosis; Venous Thromboembolism | interventions — Tinzaparin

INTERVENTIONS:
Drug: Tinzaparin sodium

SUMMARY:
The purpose of this study is to assess the long-term treatment of patients with proximal venous thrombosis through the administration of subcutaneous low-molecular-weight heparin (tinzaparin sodium) versus the standard care use of intravenous heparin followed by oral warfarin sodium.

DETAILED DESCRIPTION:
The accepted treatment for acute deep vein thrombosis (DVT) is initial continuous intravenous heparin followed by long-term oral anticoagulant therapy. Improvements in the methods of clinical trials and the use of accurate objective tests to detect venous thromboembolism have made it possible to perform a series of randomized trials to evaluate various treatments of venous thromboembolism.

The specific objectives of the Main LITE Study are:

* to determine if low-molecular-weight heparin, given subcutaneously once daily without laboratory monitoring, is more effective than adjusted oral warfarin sodium in the reduction of mortality rate.
* to determine if such a low-molecular-weight heparin therapy is more cost-effective than present standard care methods.
* to determine the incidence of Factor V Leiden and Prothrombin 20210A mutant genetic abnormalities.

ELIGIBILITY:
Inclusion Criteria:

* Patients having a first or recurrent episode of acute proximal vein thrombosis

Exclusion Criteria:

* Presence of familial bleeding diathesis or presence of active bleeding contraindicating anticoagulant therapy
* Receiving therapeutic heparin or therapeutic low-molecular-weight heparin for more than 48 hours or have already been on warfarin for more than 2 days for the treatment of proximal deep vein thrombosis
* Receiving long-term warfarin treatment
* Females who are pregnant
* Known allergy to heparin, warfarin sodium, or bisulfites
* History of heparin-associated thrombocytopenia
* Severe malignant hypertension
* Hepatic encephalopathy
* Severe renal failure
* Inability to attend follow-up due to geographic inaccessibility
* Inability or refusal to give informed consent
* Recent neurological or opthalmic surgery (within the previous 14 days)
* Pulmonary embolism requiring thrombolytic therapy, surgical thrombectomy, or vena cava interruption
* Life expectancy of less than 3 months
* Taking ASA prior to randomization and unable to discontinue this medication during the 84 day study treatment period

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 910
Dates: Start 1994-12; Study Completion 2002-03

PRIMARY OUTCOMES:
objectively documented recurrent venous thromboembolism during initial treatment or during the 12 week follow-up period
death during initial treatment or during the 12 week follow-up period
safety endpoint for assessing harm was the occurrence of bleeding (all, major or minor) during the 12 week treatment interval

SECONDARY OUTCOMES:
recurrent venous thromboembolism at 12 months
death at 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Russell D Hull, MBBS, MSc, Principal Investigator — University of Calgary
Locations (1):
- Thrombosis Research Unit, University of Calgary, Calgary, Alberta, Canada

REFERENCES:
- [Background] Koopman MM, Prandoni P, Piovella F, Ockelford PA, Brandjes DP, van der Meer J, Gallus AS, Simonneau G, Chesterman CH, Prins MH. Treatment of venous thrombosis with intravenous unfractionated heparin administered in the hospital as compared with subcutaneous low-molecular-weight heparin administered at home. The Tasman Study Group. N Engl J Med. 1996 Mar 14;334(11):682-7. doi: 10.1056/NEJM199603143341102. PMID 8594426
- [Background] Levine M, Gent M, Hirsh J, Leclerc J, Anderson D, Weitz J, Ginsberg J, Turpie AG, Demers C, Kovacs M. A comparison of low-molecular-weight heparin administered primarily at home with unfractionated heparin administered in the hospital for proximal deep-vein thrombosis. N Engl J Med. 1996 Mar 14;334(11):677-81. doi: 10.1056/NEJM199603143341101. PMID 8594425
- [Background] Lancaster TR, Singer DE, Sheehan MA, Oertel LB, Maraventano SW, Hughes RA, Kistler JP. The impact of long-term warfarin therapy on quality of life. Evidence from a randomized trial. Boston Area Anticoagulation Trial for Atrial Fibrillation Investigators. Arch Intern Med. 1991 Oct;151(10):1944-9. PMID 1929681
- [Background] Laird NM, Ware JH. Random-effects models for longitudinal data. Biometrics. 1982 Dec;38(4):963-74. PMID 7168798